CLINICAL TRIAL: NCT00802334
Title: Therapeutic Drug Monitoring of the Generic Lopinavir/Ritonavir Tablets 200/50 mg in the Thai HIV-infected Patient
Brief Title: TDM of Generic Lopinavir/Ritonavir 200/50 mg
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: The Government Pharmaceutical Organization (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 095; IRB414/50
Record Dates: First submitted 2008-05-29; First posted 2008-12-04 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV
Keywords: generic lopinavir/ritonavir; therapeutic drug monitoring; safety and efficacy
MeSH Terms: interventions — Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: generic lopinavir/ritonavir

INTERVENTIONS:
Drug: generic lopinavir/ritonavir — 1. Screening visit
     • Clinical and safety laboratory assessment. Viral load for patients on a PI-based regimen, if a VL results ≤ 3 months is not available
  2. Baseline visit
     • (Within 30 days after screening) Baseline clinical and laboratory assessment, patients who were on a Kaletra SGC formulation before baseline will undergo TDM. Start generic lopinavir/ritonavir tablets 200/50 in a 400/100mg bid dosage. Backbone will be chosen on the discretion of the study physician
  3. Week 4
     * Steady state TDM lopinavir and ritonavir, at 10-12 hr after the last intake (Cmin)
  Clinical, safety and laboratory assessment
  Week 12: Clinical, safety and efficacy laboratory assessment Week 24: Clinical, safety and efficacy laboratory assessment Week 48: Clinical, safety and efficacy laboratory assessment

SUMMARY:
Evaluating the bioavailibility safety and efficacy of the generic LPV/RTV 200/50 mg tablet formulation in a 400/100 mg BID dose in Thai HIV infected individuals.

DETAILED DESCRIPTION:
The original solid oral formulation of lopinavir/ritonavir was a soft gel capsule (SGC) in a 133/33 mg formulation. This formulation requires refrigerated storage and need to be administered with food[4]. Recently Abbott developed a new formulation of this fixed combination, a 200/50 mg tablet (Aluvia). This formulation showed to be bioequivalence to the old formulation, don't need refrigerated storage and has diminished food effect[5].

This are profound advantages for the developing world, but till now Aluvia is not available in Thailand yet, and if it will, the price might be an issue for most of the HIV-infected Thai patients.

The Indian company Matrix has produced the generic formulation of Abbott's Aluvia. In Indian healthy volunteers this tablet formulation has proven to be bioequivalent to Abbott's Aluvia in a 400/100 mg bid dosing (unpublished data). Implementing this drug in Thai clinical practice will save a huge amount of costs and, as a result, will make the second line regimen more accessible for the Thai HIV-infected population. We expect that the BE data from the Indian population can be extrapolated to the Thai population, but to confirm this and in order to register this drug in Thailand an extensive therapeutic drug monitoring (TDM) of 100 patients has to be done. To meet these regulatory criteria HIVNAT will coordinate and assess a TDM trial in Thai HIV-infected patients who are eligible for using the generic 200/50 mg lopinavir/ritonavir tablets 200/50 mg.

This is open-label, single-center phase-II trial in 100 HIV-infected subjects. Patients can be either treatment-naïve or treatment-experienced when entering this clinical trial. After meeting the in- and exclusion criteria, patients will start with lopinavir/ritonavir new formulation 400/100 mg bid with a low fat diet, plus 2 nucleoside reverse transcriptase inhibitors (NRTIs). The choice of the 2 NRTIs is at the discretion of the investigator. Only patient who are on Kaletra SGC will undergo TDM sampling at baseline. Although the paper of Klein et al. showed diminished food effect[5] we still will advice our patient to take it with food, until more data on the generic product becomes available, confirming the lack of food effect on the pharmacokinetics.

Once patients are included a (generic) lopinavir/ritonavir based regimen will be designed and initiated. Patients who were on a Kaletra SGC based regimen before baseline will undergo TDM at base line. Therapeutic drug monitoring of lopinavir will be done after 4 weeks, to ensure steady state. At baseline and week 4 safety data will be obtained.

After the first 30 patients showed good bioavailibility, the other 70 subjects will be followed up for total of 48 weeks to obtain safety and efficacy data

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Evidence of HIV infection (confirmed positive ELISA and/or documented history of measurable HIV RNA)
3. Age> 18 years
4. On a standard PI containing HAART regimen with 2 NRTIs with a VL < 50 copies for at least 12 weeks OR ARV-naive patients, or patient on a NNRTI based regimen
5. Currently having no AIDS defining illness
6. Willing to adhere to the protocol requirements

Exclusion Criteria:

1. Any history of taking CYP450 inhibitors or inducers, or any gastric acid-reducing drugs within 14 days of enrollment in the study
2. Current pregnancy or lactating
3. Active opportunistic infection
4. ALT/ AST more than 2 x upper limit
5. creatinine more than 1.5 time the upper limit
6. Relevant history or current condition, illness that might interfere with drug absorption, distribution, metabolism or excretion
7. History of sensitivity/idiosyncrasy to the drug or chemically related compounds or excipients which may be employed in the study.
8. Active drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To determine the Cmin levels of the generic lopinavir/ritonavir tablets 200/50 mg in Thai HIV-infected patients | 18 months

SECONDARY OUTCOMES:
To assess 48 weeks safety and tolerability of the generic lopinavir tablets 200/50 mg for the standard dosing regimen | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Anchalee Avihingsanon, MD, PhD, Principal Investigator — HIV-NAT, Thai Red Cross - AIDS Research Centre
Locations (1):
- HIV-NAT, Bangkok, Thailand

REFERENCES:
- [Result] Ramautarsing RA, van der Lugt J, Gorowara M, Sophonphan J, Ananworanich J, Lange JM, Burger DM, Phanuphak P, Ruxthungtham K, Avihingsanon A. Pharmacokinetics and 48-week safety and efficacy of generic lopinavir/ritonavir in Thai HIV-infected patients. Antivir Ther. 2013;18(2):249-52. doi: 10.3851/IMP2324. Epub 2012 Aug 23. PMID 22908131
- [Derived] van der Lugt J, Lange J, Avihingsanon A, Ananworanich J, Sealoo S, Burger D, Gorowara M, Phanuphak P, Ruxrungtham K. Plasma concentrations of generic lopinavir/ritonavir in HIV type-1-infected individuals. Antivir Ther. 2009;14(7):1001-4. doi: 10.3851/IMP1410. PMID 19918104
- See also: HIV-NAT's website — http://www.hivnat.org